CLINICAL TRIAL: NCT05593562
Title: A Clinical Trial to Evaluate Absorption, Metabolism and Excretion of [14C]SPH3127 in Healthy Chinese Adult Male Subjects (Human Mass Balance and Biotransformation Study of [14C]SPH3127)
Brief Title: Study on Human Mass Balance of SPH3127 Tablets
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPH3127-105
Record Dates: First submitted 2022-10-15; First posted 2022-10-25 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-10

CONDITIONS: Primary Mild and Moderate Hypertension
MeSH Terms: interventions — SPH3127

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH3127 (Experimental): Oral 100 mg [14 c] SPH3127 mixed suspension
  Interventions: Drug: SPH3127

INTERVENTIONS:
Drug: SPH3127 — Oral 100 mg [14 c] SPH3127 mixed suspension

SUMMARY:
To quantitatively analyze the total radioactivity in the excreta of healthy male subjects after oral administration of [14C] SPH3127, and determine the cumulative excretion rate and main excretion routes of radioactive substances; to investigate the partition in whole blood and plasma and the pharmacokinetics of total radioactivity in plasma after a single oral administration of [14C]SPH3127 in healthy male subjects; to identify the main metabolites in healthy male subjects after an oral administration of [14C] SPH3127, determine the main biotransformation pathways and main metabolites, quantitatively analyze the concentration of SPH3127 and main metabolites in plasma by validated LC-MS/MS method, and establish the pharmacokinetic parameters of SPH3127 and its main metabolites in plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male;
2. Age: 18-45 years (inclusive);
3. Body weight: the body weight of the subject is ≥ 50 kg, and the body mass index (BMI) is between 19 and 26 kg/m2 (inclusive);
4. Subject who fully understands the objective, requirements, content, process and possible adverse reactions of this trial, volunteers for the trial, is able to complete the trial according to the trial requirements and comply with study instructions, and the process of obtaining informed consent conforms to GCP;
5. Subject who can communicate well with the investigator and complete the trial according to the protocol.

Exclusion Criteria:

1. Those with clinically significant abnormalities in physical examination, vital signs, laboratory tests, thyroid function, 12-lead ECG, chest CT, abdominal ultrasound and other examinations;
2. Those positive for combined detection of hepatitis B surface antigen or e antigen, hepatitis C virus antibody IgG, human immunodeficiency virus antigen/antibody and Treponema pallidum antibody;
3. Screening for SARS-COV-2 infection: those with clinically significant abnormalities in C-reactive protein or positive for SARS-COV-2 RNA;
4. Those who have used any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 30 days prior to screening;
5. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements within 14 days prior to screening;
6. Those who have a history of any clinical serious disease or any disease or condition that the investigator thinks may affect the trial results, including but not limited to the medical history of circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic disorders;
7. Those with a personal history or family history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmias, torsades de pointes, ventricular tachycardia, atrioventricular block, prolonged QT syndrome;
8. Those who have undergone major surgery or have incomplete healing of surgical incision within 6 months prior to screening; major surgery includes, but is not limited to, any surgery with significant bleeding risk, prolonged general anesthesia, or open biopsy or significant traumatic injury;
9. Those with allergic constitution, such as a known history of allergy to two or more substances; or those who, at the investigator's discretion, may be allergic to the investigational drug or its excipients;
10. Those with perianal disease, irritable bowel syndrome, inflammatory bowel disease with regular/ongoing hematochezia;
11. Those with habitual constipation or diarrhea;
12. Those who drink excessively or drink frequently within 6 months prior to screening, that is, drinking more than 14 units of alcohol every week and unable to quit during the trial; or the alcohol breath test result is > 0 mg/dL during screening period;
13. Those who smoke more than 5 cigarettes a day or habitually used nicotine-containing products within three months prior to screening, and are unable to quit during the trial;
14. Those who have a history of drug abuse within 3 months prior to screening or have a positive urine test for illegal drugs during screening;
15. Those who habitually drink grapefruit juice or excessive tea, coffee and/or caffeinated drinks, and are unable to quit during the trial;
16. Those who need to be exposed to radioactive conditions for a long time; or those who have had significant radiation exposure or participated in radiopharmaceutical labeling test within 1 year prior to screening;
17. Those who have a history of fear of needles or blood fainting, and who have difficulty in blood collection or are unable to tolerate venous puncture for blood collection;
18. Those who have participated in any other clinical trial within 3 months prior to screening;
19. Those who have been vaccinated within one month prior to screening or who plan to be vaccinated during the trial;
20. Those who have fertility or sperm donation plans during the trial and within one year after the completion of the trial, or do not agree to take strict contraceptive measures with their female partners throughout the trial and for up to one year after the completion of the trial;
21. Those who have lost blood or donated blood up to 200 mL within 3 months or have received blood transfusion within 1 month prior to screening;
22. Subjects who are considered by the investigator as having any factors unsuitable for this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion rate of total radioactive substances in excreta | 240 hours
  Cumulative excretion rate of total radioactive substances in excreta(urine and faeces).
The concentration of SPH3127 in plasma | Sampling performed at predose, and 10 minute,20 minute,0.5, 0.75, 1, 1.5, 2, 4, 8, 12, 24,48,72,96,120,144and 168 hours post-dose.
  The concentration of SPH3127 in plasma was determined by liquid chromatography tandem mass spectrometry (LC-MS/MS).
The total radioactivity in the collected plasma samples | up to 168 hours
  The total radioactivity in the collected plasma samples was measured directly by liquid scintillation counter.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Predose and 240 hours post-dose.
  Adverse event type, incidence, correlation with study drug

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China